CLINICAL TRIAL: NCT06437574
Title: Lowering Cholesterol in Prostate Cancer to Target Rapamycin-Insensitive Companion of MTOR (TORC2) in T-Cell Surface Glycoprotein CD8 Alpha Chain (CD8+) Lymphocytes
Brief Title: Intensive Cholesterol-Lowering and CD8+ T Cells in Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Hyung L. Kim, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003290; R01CA280060 (NIH)
Record Dates: First submitted 2024-05-23; First posted 2024-05-31 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ezetimibe, Simvastatin Drug Combination; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intensive Lipid Lowering (Experimental): Single arm with dual agents (ezetimibe and simvastatin) or single agent (ezetimibe). These agents target the two primary sources of cholesterol, absorption in the gut (ezetimibe) and synthesis in the liver (simvastatin). The dual agents are available in a single pill that is FDA approved and sold under the trade name, Vytorin.
  Interventions: Drug: Vytorin; Drug: Ezetimibe

INTERVENTIONS:
Drug: Vytorin — Vytorin is a drug combination (Ezetimibe and Simvastatin) that targets the two primary sources of cholesterol, absorption in the gut and synthesis in the liver.
Drug: Ezetimibe — Ezetimibe is a drug that targets one of the primary sources of cholesterol, absorption in the gut.

SUMMARY:
To test the hypothesis that intensive cholesterol lowering (iCL) therapy has anti-tumor immune modulating activity, the investigators will conduct an open-label, single-arm phase II trial in prostate cancer patients who are in active surveillance and undergoing a planned surveillance biopsy in 3-6 months. Eligible patients will initiate iCL with Vytorin®(group 1, 2, and 3), an FDA-approved combination of ezetimibe and simvastatin used to lower atherogenic low density lipoprotein cholesterol (LDL-C) or Ezetimibe (group 4). Starting dose will be determined by current statin use and LDL-C levels. Dose modifications of VYTORIN will be employed with the goal of achieving LDL-C <70 mg/dl. Dose adjustment is not allowed for ezetimibe.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. At least one Atherosclerotic Cardiovascular Disease (ASCVD) risk factor, such as:

   1. ≥ 50 years of age
   2. Hypertension
   3. Hypercholesterolemia
   4. Diabetes
   5. Current or former smoker
   6. First-degree family history of any cardiovascular heart disease
   7. BMI > 25
   8. On hypertension treatment, statin, and/or aspirin therapy
4. Patients with clinically localized prostate cancer. That is Low or intermediate risk prostate cancer deﬁned as:

   1. Pre-operative PSA (Prostate Specific Antigen) ≤ 20.0 ng/ml
   2. Clinical stage T1c or cT2
   3. Gleason score 3+3 or 3+4 or 4+3
5. Patients on AS with plans for surveillance biopsy
6. No previous treatment for prostate cancer with radiotherapy, chemotherapy, or hormonal therapy
7. Ability to take oral medication and be willing to adhere to once daily, oral Vytorin or ezetimibe.
8. Agree to avoid consumption of grapefruit and grapefruit juice ≥ one quart per day throughout study duration.

Exclusion Criteria:

1. Current use of medications contraindicated for use with a statin such as strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, posaconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, and nefazodone).
2. Current use of medications contraindicated for use with ezetimibe (i.e., gemfibrozil, cyclosporine, or danazol).
3. History of allergic or severe reaction to a either study agent.
4. History of moderate or severe myalgia with statin use.
5. Acute liver failure or decompensated cirrhosis
6. Already on maximum VYTORIN dose (10/80)
7. Already on medication(s) known to interact with Vytorin or Ezetimibe that may prevent protocol-based escalation of cholesterol-lowering therapy from pre-enrollment baseline.
8. Already on a PCSK9 inhibitor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Pre/Post-change in percent prostate infiltrating CD8+ T lymphocytes. | 3 to 6 months of cholesterol-lowering intervention
  Our primary hypothesis is that maximum cholesterol lowering will increase CD8+ memory T cells and increase CD8+ T cell infiltration into prostate tissue. Change in CD8+ T cells in the prostate from baseline to 3 to 6 months is the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Kim, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No